CLINICAL TRIAL: NCT02423174
Title: Evaluation of Safety and Effectiveness of the FMwand Ferromagnetic Surgical System During Total Mesorectal Excision Surgery
Brief Title: Eval. of Safety and Effectiveness of the FMwand Ferromagnetic Surgical System During Total Mesorectal Excision Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Funding
Sponsor: Domain Surgical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FMW-IT-02
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total Mesorectal Excision: Patients with an indication for surgical intervention for a total mesorectal excision
  Interventions: Procedure: Total Mesorectal Excision; Device: FMwand Surgical System

INTERVENTIONS:
Procedure: Total Mesorectal Excision — Surgical intervention with the FMwand Surgical System
Device: FMwand Surgical System

SUMMARY:
The objective of the clinical trial is to determine the suitability of the FMwand Ferromagnetic Surgical System for Total Mesorectal Excision Surgery.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed rectal cancer to the lower two-thirds of the rectum (higher and T2 N0 or N+)
* Amenable for standard surgery procedures using electrocautery, argon beam, lasers or other conventional tissue removal modalities
* ECOG status ≤ 2
* Life expectancy >3 months
* Age ≥ 18 years old
* Age ≤ 80 years old
* Ability to provide written informed consent and HIPAA forms prior to admission to this study
* Willingness to meet all of the expected requirements of this clinical protocol

Exclusion Criteria:

* Patient with metastasis
* History of radiotherapy or chemotherapy for the treatment of rectal cancer
* Uremia - BUN>40
* Hemodialysis
* Existing urinary or fecal incontinence
* Pregnant or lactating
* Previously diagnosed coagulopathy or bleeding diathesis
* Currently, or within the previous 10 days prior to surgery, taking any medications that would produce bleeding diathesis including but not limited to, Plavix, warfarin, NSAIDs, clopidogrel, ticlopidine or valproic acid
* History of significant cardiac disorders that would necessitate special fluid management protocols
* History of acute myocardial infarction and/or acute angina
* INR >1.4 in the 24 hours prior to surgery
* PTT >40 in the 24 hours prior to surgery
* Platelet count <100K in the 24 hours prior to surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for surgical intervention for a total mesorectal excision
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Serious Adverse Events as a Measure of Safety and Feasibility | 1 day after surgery
  Safety and feasibility will be assessed by evaluating intra-operative serious adverse events, if any, and their relationship with the FMwand Ferromagnetic Surgical System

SECONDARY OUTCOMES:
Post-operative Drainage | Beginning day 2 after surgery and for the duration of the hospital stay, an expected average of 6 days
  Volume of drainage and drain residence time
Onset of urinary or fecal incontinence | Beginning day 2 after surgery and for the duration of the hospital stay, an expected average of 6 days
  Incidence of urinary or fecal incontinence attributed to post-surgical nerve dysfunction
Duration of Procedure | During Procedure
  Total operative time
Duration of TME resection | During procedure
  Total resection time
Evaluation of post-operative complications | 12 weeks after surgery
  Evaluation of pelvic fibrosis, adherences, abscess or fluid collections assessed by CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Izzo, MD, Principal Investigator — Istituto Nationale Tumori IRCCS - Fondazione "G Pascale"

REFERENCES:
- [Background] Bowers CA, Burns G, Salzman KL, McGill LD, Macdonald JD. Comparison of tissue effects in rabbit muscle of surgical dissection devices. Int J Surg. 2014;12(3):219-23. doi: 10.1016/j.ijsu.2013.12.014. Epub 2014 Jan 7. PMID 24406264
- [Background] MacDonald JD, Bowers CA, Chin SS, Burns G. Comparison of the effects of surgical dissection devices on the rabbit liver. Surg Today. 2014 Jun;44(6):1116-22. doi: 10.1007/s00595-013-0712-4. Epub 2013 Sep 5. PMID 24006128
- [Background] Tok, S et al. Comparison of a Novel Thermal Surgical Technology with Monopolar and Carbon Dioxide Laser in a Rat Glioma Model. Poster presentation.